CLINICAL TRIAL: NCT04549818
Title: Does Sacral Neuromodulation Relieve Chronic Pelvic Cancer Pain, Compared With Medical Treatment?
Brief Title: Analgesic Efficacy of Sacral Neuromodulation for Pelvic Cancer Pain: A Preliminary Report
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Diab Fuad Hetta, anesthesia dep. south egypt cancer institute, El methaque st., assuit city, Egypt, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SECI2020
Record Dates: First submitted 2020-08-31; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sacral neuromodulation (Experimental): Sacral neuromodulation group, will be treated with Stimulation of the sacral nerve roots by placement of a lead and generator, typically using an implanted InterStim® device that provides constant electrical stimulation to the S 2, 3 and 4 nerve roots, for 2-week trial stimulation
  Interventions: Device: sacral neuromodulation
- medical therapy (No Intervention): this group will be treated with sustained release morphine tablets for pain control

INTERVENTIONS:
Device: sacral neuromodulation — Sacral neuromodulation group, N=22 will be treated with Stimulation of the sacral nerve roots by placement of a lead and generator, typically using an implanted InterStim® device that provides constant electrical stimulation to the S 2, 3 and 4 nerve roots, for 2-week trial stimulation
  Arms: sacral neuromodulation

SUMMARY:
in this trial, we will test the analgesic efficacy of sacral neuromodulation for patients with pelvic cancer, complaining of chronic pelvic pain in comparison to medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age, 18-70
* Pain localized to the pelvic and perineal region
* The pain is due to pelvic cancer or chronic pelvic pain after pelvic surgery for cancer
* The intensity of pain assessed by VAS (visual analogue pain scale) > 7
* Importantly, the included participants should gain > 50% reduction of their pain in response to sacral roots block, S2,3 and 4 with bupivacaine 0.5%, 2 ml for each root

Exclusion Criteria:

* Coagulopathy
* Infection at site of maneuver
* Abnormal Psychological behavior that interfere with integrity of obtained data

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-09-10 (Estimated); Primary Completion 2021-09-10 (Estimated); Study Completion 2021-12-10 (Estimated)

PRIMARY OUTCOMES:
The change of intensity of pain | The outcome will be measured at day 15 postoperatively.
  The intensity of pain measured by VAS pain score (visual analogue pain scale) where 0= no pain and 10=the maximum tolerated pain